CLINICAL TRIAL: NCT05011968
Title: Intervention Study With Crop Lettuce Enriched With Iodine
Brief Title: Intervention Study on Iodine Biofortification Vegetables ( Nutri-I-Food
Acronym: Nutri-I-Food
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Sonya Vasto, Associate professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nutr-I-Food2019
Record Dates: First submitted 2021-07-18; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Healthy Individuals
Keywords: functional food; biocarrier; Iodine
MeSH Terms: interventions — Iodine

STUDY DESIGN:
Intervention Model Description: The study were designed by two cohorts The control group and the interventional group. The intervention lasted for 10 days and 100gr of lettuce per day was consumed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: (control group) (Experimental): The control group was assigned to crop lettuce without any biofortification but with the same characteristic of bioforticated lettuce (soil, water, harvesting time)
  Interventions: Dietary Supplement: Lettuce with not biofortification
- Experimental: intervention group (Experimental): The intervention group was assigned to biofortificated Iodine crop lettuce.
  Interventions: Dietary Supplement: Lettuce biofortificated with Iodine

INTERVENTIONS:
Dietary Supplement: Lettuce with not biofortification — Lettuce without any biofortification was assigned to each participant belonging to the control group which ate 100gr every day for 10 days
  Arms: No Intervention: (control group)
Dietary Supplement: Lettuce biofortificated with Iodine — Lettuce with Iodine biofortification was assigned to each participant belonging to the intervention group which ate 100gr every day for 10 days
  Arms: Experimental: intervention group

SUMMARY:
The aim of the project is to study of the influence of Lettuce crop enriched with Iodine on Thyroid hormone synthesis. Secondary outcome to find out iodine presence in urine in order to evaluate vegetables, like little crop, as Iodine biocarrier

DETAILED DESCRIPTION:
Several human pathologies are caused by deficiencies of some mineral elements. These deficiencies can be overcome through careful dietary diversification and mineral supplementation. An alternative or even complementary way is represented by the intake of bio-fortified foods. In the field of mineral deficiency increasing the bioavailable mineral concentration in vegetables intended for human consumption; can be a useful tool to prevent many harmful pathologies. Therefore, in this scenario, it appears very important to identify the right dosages and the most effective methods of administration to bio-fortify vegetables with a strong nutritional-health connotation.

The present project aim to investigate the benefits of fortified food intake in a cohort of healthy individuals. Specifically, healthy individuals received lettuce enriched with iodine and after 10 days plasma and urine samples were collected . Each subject was subjected to two venous blood samples taken at the beginning of the observation and at the end (after 10 days). The samples thus obtained were transported in certified containers for the safe transport of biological samples, and, subsequently, processed by the laboratories of the Molecular Biology section of the University of Palermo. Serum and plasma will be obtained from each blood sample. All information thus obtained will be recorded in a database in which each person will be identified with a numerical code, in order to comply with current privacy regulations. Body weight, Barefoot standing height, Body mass index, Body composition will be measured in the different groups of study. Samples will be analyzed and compared for glucose, albumin, total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, uric acid, creatinine, AST, ALT, γ-GT, ALP, bilirubin, Ferritin, free Iron, transferrin, total proteins, Magnesium, Calcium, insulin, osteocalcin,TSH, FT3, FT4, hematocrit, hs-CRP, Bone metabolism (Osteocalcin, parathyroid hormone, CTX, Calcitonin), Vitamin D Calcium, Phosphate, Potassium, gastric hormones ( GIP, GLP1, GLP2, ghrelin, glucagon, PYY, CCK) oxidative stress markers (LDL-ox, AGE, urinary 8-iso-prostaglandin F (PGF)2alpha) and inflammatory markers(IL-1, TNF, IL-6, IL-10)

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* age: 18-65 years
* healthy status
* no drug therapy or integration therapy

Exclusion Criteria:

* Inflammatory chronic disease
* use of medication or suffering from any condition
* pregnancy
* breastfeeding
* current smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Serum Thyroid markers | 10 days
  serum levels of free tri-iodothyronine (FT3 ng/L), free thyroxine (FT4 ng/L) and thyroid-stimulating hormone (TSH ng/L) will be assessed at baseline and after 10 days
Urine Iodine concentration | 10 days
  Urine Iodine concentration (mg/l) will be assessed at baseline and after 10 days
Haematology and serum chemistry values 1 | 10 days
  glucose (mg/dL), albumin( mg/dL), total cholesterol (mg/dL), HDL-cholesterol (mg/dL), LDL-cholesterol (mg/dL), triglycerides(mg/dL), uric acid(mg/dL), creatinine(mg/dL) will be assessed at baseline and after 10 days
Haematology and serum chemistry values 2 | 10 days
  insulin (mUI/L) will be assessed at baseline and after 10 days
Haematology and serum chemistry values 3 | 10 days
  Potassium (mmol/L) will be assessed at baseline and after 10 days
Haematology and serum chemistry values 4 | 10 days
  Ferritin (mg/L), free Iron (mg/L), transferrin (mg/L), total proteins (mg/L), Magnesium (mg/L), Calcium (mg/L), Vitamin D (mg/L), HCRP (mg/L), Phosphate (mg/L), Cortisol (mg/L)will be assessed at baseline and after 10 days
Haematology and serum chemistry values 5 | 10 days
  AST (U/L), ALT (U/L), γ-GT(U/L), ALP(U/L) will be assessed at baseline and after 10 days

SECONDARY OUTCOMES:
body mass index (BMI) | 10 days
  BMI (kg/m2) All these measurements will be assessed at baseline and after 10 days
body composition (%) | 10 days
  lean mass as percent of body weight and fat mass as percent of body weight will be assessed at baseline and after 10 days
Gastric Hormones | 10 days
  GIP (pg/m), GLP1 (pg/m), GLP2 (pg/m), ghrelin (pg/m), glucagon (pg/m), PYY (pg/m), CCK(pg/m) measured in plasma will be assessed at baseline and after 10 days
Oxidative stress markes | 10 days
  LDL-ox (ug/mL), AGE(ng/mL), urinary 8-iso-prostaglandin F (PGF)2alpha (ng/mL) will be assessed at baseline and after 10 days
Bone metabolism | 10 days
  Osteocalcin(ng/L), parathyroid hormone (ng/L), CTX, Calcitonin (ng/L) measured in plasma will be assessed at baseline and after 10 days
Inflammatory markers | 10 days
  IL-1 (pg/mL), TNF(pg/mL), IL-6(pg/mL), IL-10(pg/mL) measured in plasma will be assessed at baseline and after 10 days
Weigh | 10 days
  Weight (Kg) will be assessed at baseline and after 10 days
Hight | 10 days
  Hight (m) will be assessed at baseline and after 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Vasto, PhD, Principal Investigator — D. Biological, Chemical and Pharmaceutical Sciences and Technologies, Palermo University
Locations (1):
- Department of Biological, Chemical and Pharmaceutical Sciences and Technologies, Palermo University, Palermo, Italy